CLINICAL TRIAL: NCT05504187
Title: An Open-label, Phase 2 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of KP104 in Subjects With Thrombotic Microangiopathy Secondary to Systemic Lupus Erythematosus
Brief Title: Study to Evaluate Safety, Tolerability and Pharmacodynamics of KP104 in Participants With Thrombotic Microangiopathy Secondary to Systemic Lupus Erythematosus
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kira Pharmacenticals (US), LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KP104-202
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic lupus erythematosus; Thrombotic microangiopathy; Dose Selection; Proof of Concept; KP-104
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Thrombotic Microangiopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part 1: Dose Optimization Cohort 1, Dose 1 (Experimental): Participants will be administered with KP104 as a weekly maintenance dose for 24 Weeks. After the last participant completes 6 weeks of treatment, all available data, including safety, PK, PD, and modeling results, will be reviewed by the Internal Data Review Committee (IDRC) to determine Dosing Regimen 2
  Interventions: Drug: KP104
- Part 1: Dose Optimization Cohort 2, Dose 2 (Experimental): Participants will be administered with KP104 dose regimen 2 for 24 Weeks. After the last participant completes 6 weeks of treatment, all available data, including safety, PK, PD, and modeling results, will be reviewed by the IDRC to determine Dosing Regimen 3.
  Interventions: Drug: KP104
- Part 1: Dose Optimization Cohort 3, Dose 3 (Experimental): Participants will be administered with KP104 dose regimen 3 for 24 Weeks. After the last participant completes 6 weeks of treatment, all available data, including safety, PK, PD, and modeling results, will be reviewed by IDRC to determine the Optimal biologic dose (OBD) for Part 2.
  Interventions: Drug: KP104
- Part 2: OBD Cohort, Dose 4 (Experimental): Participants will be administered with KP104 OBD for 24 Weeks.
  Interventions: Drug: KP104

INTERVENTIONS:
Drug: KP104 — KP104 will be administered.

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and efficacy of KP104 in participants with systemic lupus erythematosus (SLE)-Thrombotic microangiopathy (TMA). The study consists of 2 parts: Part 1 (Dose Optimization) and Part 2 (Proof of Concept). All participants will receive KP104 in combination with standard of care (SOC) for SLE-TMA.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for SLE per the 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) criteria.
* Decrease in platelet count to less than (<)150,000/microliters (mcL).
* Abnormal renal function.
* Females of childbearing potential with negative pregnancy test and males must agree to practice effective contraception from Screening until 28 days after the End of study (EOS) visit.
* Willing and able to provide informed consent.
* Evidence of microangiopathic hemolytic anemia

Exclusion Criteria:

* Diagnosis of other TMA syndromes.
* A renal biopsy within 7 days of screening that shows exclusively chronic changes of TMA.
* Positive Coombs test at the time of TMA diagnosis.
* Active or unresolved Neisseria meningitidis infection at screening.

Only key inclusion and exclusion criteria have been included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Parts 1 and 2: Number of participants with Treatment-emergent adverse events (TEAEs), treatment-emergent serious adverse events (TESAEs) and Adverse events of special interest (AESIs) | Up to 24 weeks
Part 2: Percent change from Baseline in platelet count | Baseline (Day 1) and up to Week 12
Part 2: Percent change from Baseline in serum lactate dehydrogenase (LDH) levels | Baseline (Day 1) and up to Week 12

IPD SHARING:
Plan to Share IPD: Yes